CLINICAL TRIAL: NCT05852002
Title: A Clinical Study of 35 kDa Hyaluronan Fragment in Treatment of Pain and Discomfort Associated With Advanced Lung Cancer
Brief Title: A Clinical Study of Pain and Discomfort Associated With Advanced Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhia Impex LLC (Industry)
Collaborators: Mongolian National University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSHN004
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-04

CONDITIONS: Advanced Lung Cancer
Keywords: 35kDa hyaluronan fragment; palliative care; pain and discomfort; cough; fatigue
MeSH Terms: conditions — Pain; Cough; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 35 kDa hyaluronan fragment injection (Experimental): 35kDa hyaluronan fragment was produced by using hyaluronidase PH20 to cleave 1600kDa hyaluronan ( HA1600 ). Batch number of 35 kDa hyaluronan fragment injection is L20200708MP07707,and the injection was approved by Ministry of Health, Mongolia.
  Interventions: Drug: 35 kDa hyaluronan fragment

INTERVENTIONS:
Drug: 35 kDa hyaluronan fragment — 100 mg of 35kDa hyaluronan fragment was injected deeply into abdominal fat layer once a day for 28 consecutive days.
  Other Names: B-HA

SUMMARY:
In this research, the patients with advanced lung cancer accompanied by pain and discomfort were treated by injecting freshly manufactured tissue permeable hyaluronan fragment HA35 into the tissue under abdominal adipose.

DETAILED DESCRIPTION:
Pain is generally considered the most common symptom of lung cancer. The three most common causes of pain in patients with advanced lung cancer are: 1. metastasis of lung cancer to the bones, which accounts for approximately 34 percent of lung cancer pain; 2. Presence of a Pancoast tumor, located at the top of the lung close to the brachial plexus nerves and cervical sympathetic nerves, which accounts for approximately 31 percent of lung cancer pain; 3. Spread of the cancer into the chest wall, accounting for approximately 21 percent of lung cancer pain.

Palliative care is a specialized field that aims to alleviate symptoms and maximize the patient's quality of life. Palliative care does not focus on curing the disease or prolonging life, which is the goal of other cancer treatments, such as chemotherapy. However, palliative care is an important part of the patient's treatment plan and encompasses physical symptoms, psychosocial distress, spiritual distress, and caregiver distress.

The management of pain due to lung cancer may include a combination of medications, such as non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroids, opioids (pain medications), and antidepressants. For metastases to the bone, radiation therapy and the use of bisphosphonates (drugs to help prevent bone breakdown) can alleviate pain. In addition, smoking cessation (stopping smoking) is recommended, as surveys have revealed that lung cancer patients who continue to smoke after diagnosis have a higher incidence of pain and other lung cancer complications than nonsmokers and those who quit smoking.

While pain is the most common symptom of lung cancer, other symptoms include: persistent coughing，wheezing，shortness of breath，hoarseness，weight loss，loss of appetite，fatigue or feeling weak and respiratory infections (like bronchitis or pneumonia) that don't go away or keep returning.

Hyaluronidase PH20 produced 35 kDa tissue permeable low molecular weight hyaluronan fragment by cutting high molecular hyaluronan. The previous clinical studies had shown that local injection of 35 kDa hyaluronan fragment effectively relieved inflammatory pain and neuropathic pain and promoted chronic wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years old
* Sign the informed consent form voluntarily.
* Expected survival ≥3 months.
* Pathologically confirmed locally advanced, metastatic or recurrent non-small cell lung cancer (NSCLC), which is currently not suitable for local treatment such as radical surgery or radiotherapy.
* The subject has good compliance and cooperates with the follow-up.

Exclusion Criteria:

* Subjects who are receiving systematic steroid treatments before the first cell treatment.
* Subjects with a history of mental disorders or drug abuse that may influence treatment compliance.
* Women in pregnancy or lactation or are expected to be pregnant during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
A pain scale | twenty eight days
  0 represents no pain or discomfort , while 10 represents the most serious pain or discomfort.
Respiratory symptom cough | twenty eight days
  A modified pain scale was used to assess respiratory symptom cough associated with advanced lung cancer. 0 represents no cough while 10 represents the most severe cough.
Fatigue | twenty eight days
  A modified pain scale was used to assess fatigue associated with advanced lung cancer. 0 represents no fatigue while 10 represents the most severe fatigue.
The degree of facial skin brightness and facial expression or spirit | twenty eight days
  A modified pain scale was used to assess the degree of facial skin brightness and facial expression or spirit associated associated with advanced lung cancer. 0 represents the best degree of facial skin brightness while 10 represents the worst degree of facial skin brightness; 0 represents the best degree of facial expression or spirit while 10 represents the worst degree of facial expression or spirit.
chest CT scans | 3 months
  namely "significant reduction" or "significant increase" or "no significant changes" in lung tumor mass.

CONTACTS AND LOCATIONS:
Locations (1):
- Mongolian National University of Medical Sciences, Ulaanbaatar, Mongolia